CLINICAL TRIAL: NCT05250297
Title: Pregnant Women's Intention and Behavioral Regarding Cross-Trimester Regular Exercise-Based on the Theory of Planned Behavior
Brief Title: Physical Activity and Symptom Disturbance Regarding Cross-Trimester
Status: Completed | Type: Observational
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, the Office of Research and Development, Mackay Medical College
Other Study IDs: LCF-MMC107
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — standard prenatal care

SUMMARY:
This study will explore pregnant women's regular exercise intentions and behavior across trimesters (from first trimester, second trimester to third trimester).

DETAILED DESCRIPTION:
Based on the TPB, this study will explore pregnant women's regular exercise intentions and behavior across trimesters (from first trimester, second trimester to third trimester). Moreover, the study will explore the effect factors, predictors and transition factors regarding pregnant women's regular exercise intention and behavior across trimesters.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were women in 8-16 weeks of gestation with a singleton pregnancy who had no obstetric or medical complications

Exclusion Criteria:

* Excluded were those who had American college of Obstetrics and Gynecology (ACOG) absolutely contraindication exercise, such as insulin-dependent diabetes, gestational diabetes, hypertension, and multiple-gestation pregnancies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants were recruited from the prenatal outpatient departments of hospitals in Taipei, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change of physical activity across different trimesters of pregnancy | The data were collected before the intervention to childbirth: <16 week gestation, second trimester (24-28 weeks), third trimester (>36 weeks)
  The pregnancy physical activity questionnaire (PPAQ) was used to measure women's physical activity during pregnancy
Change of symptom distress across different trimesters of pregnancy | The data were collected before the intervention to childbirth: <16 week gestation, second trimester (24-28 weeks), third trimester (>36 weeks)
  The pregnancy-related symptom Disturbance was used to measure women's symptom disturbance. The highest total score was severe levels of pregnancy-related distress.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Fang Lee, PhD, Principal Investigator — Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan